CLINICAL TRIAL: NCT06414356
Title: The Effect of Outpatient Ketamine Infusion on Chronic Neuropathic Pain and PTSD: A Prospective Randomized Design
Brief Title: The Effect of Outpatient Ketamine Infusion on Chronic Neuropathic Pain and PTSD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Margaux M. Salas, PhD (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Margaux M. Salas, PhD, Senior Scientist Expert, Brooke Army Medical Center
Organization: Brooke Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 954942
Record Dates: First submitted 2024-04-29; First posted 2024-05-16 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Neuropathic Pain; PTSD
Keywords: Ketamine Hydrochloride
MeSH Terms: conditions — Neuralgia; Stress Disorders, Post-Traumatic | interventions — Ketamine; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: (1) Moderate-dose ketamine (0.50 mg/kg/hr) (Orhurhu et al., 2019), and (2) moderate-dose ketamine in combination with magnesium (750 mg/hr) (Urits et al., 2021) and (3) magnesium control (750mg/hr) will be assessed. Of note, we are adapting a delayed control treatment group design. The control group (Mg only control) will be randomly assigned to one of the treatment groups (moderate dose ketamine, or moderate dose ketamine +Mg) after 2 weeks and complete the full infusion treatment regime of the randomly selected treatment group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Moderate Dose Ketamine (Experimental): 0.5 mg/kg/hr The total amount of ketamine for each participant is dependent on their body weight in kg per ideal body weight (IBW) formula.
  This total ketamine dose will be injected into one 250 ml normal saline 0.9% solution with a rate of 62.5 ml/hr over four hours or until the contents of the bag are infused and flushed with 20 ml of normal saline
  Interventions: Drug: Ketamine
- Moderate dose ketamine + magnesium sulfate (Experimental): 0.50 mg/kg/hr ketamine + 750 mg/hr Mg
  Interventions: Drug: Ketamine + Magnesium sulfate
- Magnesium sulfate (Active Comparator): 750 mg/hr
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Ketamine — Ketamine will be placed in 250 mL normal saline and infused at a rate of 62.5 mL/hr. Participants will receive intravenous infusions of ketamine for 4 hours each day in diminishing number of dosing events per week for the full 24-week infusion regime in an outpatient setting. (ketamine 0.5 mg/kg IBW/hr)
  Other Names: Ketalar
  Arms: Moderate Dose Ketamine
Drug: Magnesium sulfate — Magnesium sulfate 3 grams will be diluted into 250 mL normal saline and infused at a rate of 62.5 mL/hr (over 4 hours until the entire contents are infused and then flushed with 20 mL of normal saline). The Mg only group will be randomly assigned to one of the treatment groups (moderate dose ketamine, or moderate dose ketamine +Mg) after 2 weeks and complete the full 24-week infusion treatment regime of the randomly selected treatment group in an outpatient setting.
  Arms: Magnesium sulfate
Drug: Ketamine + Magnesium sulfate — Participants will receive intravenous infusions of ketamine and magnesium sulfate in combination. Ketamine will be placed in 250 mL normal saline and infused at a rate of 62.5 mL/hr Participants will receive intravenous infusions of ketamine and magnesium sulfate for 4 hours each day in diminishing number of dosing events per week for the full 24-week infusion regime in an outpatient setting. (Ketamine 0.5 mg/kg IBW/hr + magnesium sulfate 3 grams diluted into 250 mL normal saline)
  Other Names: ketalar + Magnesium Sulfate
  Arms: Moderate dose ketamine + magnesium sulfate

SUMMARY:
This study is aimed to evaluate outpatient ketamine infusion within a military chronic neuropathic pain population and its effect on PTSD. Currently, this is a pilot study with 30 participants. Participants will be randomized to (1) a moderate dose ketamine, (2) moderate dose ketamine +Mg, or (3) a magnesium control group. Participants will complete self-reported pain and PTSD questionnaires throughout the ~24-week study period. The outlined strategy will provide evidence for the utility of ketamine in neuropathic pain management and pain associated comorbidities within a military population.

DETAILED DESCRIPTION:
Subjects will be recruited with no target toward ethnicity, gender, or race. Active duty, veteran, retiree, and military dependents between the ages of 18-70 years old with an established diagnosis of chronic neuropathic pain will be identified and screened for study inclusion. Enrollees will have had neuropathic pain >3 months duration, report a pain score between 4-7, and meet inclusion/exclusion criteria for the study. Since ketamine's influence on PTSD is a secondary measure, any patients with a PCL-5 score > 33 will be noted. After informed consent is obtained participants will be randomized into a (1) moderate dose ketamine, (2) moderate dose ketamine +Mg, or (3) a magnesium control group. The magnesium-only group will be randomly assigned to one of the treatment groups (moderate dose ketamine or moderate dose ketamine +Mg) after 2 weeks and complete the full infusion treatment regime of the randomly selected treatment group. Administration of ketamine will occur in diminishing number of dosing events: Week 1 & 2 will consist of 3 treatments per week. Weeks 3 & 4 will consist of 2 treatments per week. Weeks 5 & 6 will consist of 1 treatment per week. Booster treatments will be administered week 10 and week 24. Booster treatments will only be 1 infusion that week. Participants will fill out questionnaires before and after each infusion- day concerning their pain, PTSD, anxiety, depression, and quality of life. Participants will be evaluated at least 5 days prior to the first treatment and 30-35 days after the final infusion. Participants will continue their current pain management regimen during the study and be instructed to use analgesics only as needed. Pain medication use will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old with Chronic Neuropathic Pain >= 3 months
* Biologic male or biologic female
* Women of childbearing age will be included if there are no plans of pregnancy within the study period, the participant agrees to actively utilize contraception throughout the study, and agrees to pregnancy tests
* Active Duty, Veterans, and retirees
* Ketamine naïve for 1 year
* Moderate Neuropathic pain Scale 4-7

Exclusion Criteria:

* Cognitive dysfunction
* Psychiatric illness involving psychosis
* Neurocognitive disorder
* Patients with Traumatic Brain Injury (TBI)
* Acute cardiovascular disease or poorly controlled hypertension
* Untreated or uncontrolled thyroid disease
* Hyperthyroidism
* Severe liver or renal disease
* Renal impairment
* History of recent heart attack, vascular disease, or any other medical condition that may be deemed by a provider as a contraindication to receiving ketamine
* Active substance abuse
* Pregnant or lactating
* Patients who are planning to become pregnant within 12 weeks of treatment completion
* Elevated Blood Pressure/hypertension
* Known hypersensitivity to Ketamine
* Hemodynamic instability
* Respiratory depression
* Use of Theophylline or Aminophylline, Sympathomimetics and Vasopressin,
* Use of Benzodiazepines
* A history of drug abuse or dependence
* Active risk of substance use
* Patients who are not able to abide by the pre-treatment and posttreatment clinical protocol, such as food intake, abstaining from certain medications, unable to remain in the clinic for a minimum of 1 hour for observation, and cannot provide the name and phone number of the party who will pick them up post-treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Defense and Veterans Pain Rating Score (DVPRS) | Up to 32 weeks
  The DVPRS is a self-report instrument used to assess pain intensity in military personnel, veterans, and other military populations. It was specifically developed for individuals with military backgrounds and is often used in clinical settings to monitor pain levels and treatment effectiveness.
  The DVPRS consists of a Numeric Rating Scale (NRS) from 0 to 10, where 0 represents "no pain" and 10 represents "worst possible pain." Respondents rate their pain intensity by selecting the number that best corresponds to their current level of pain.
  The DVPRS questionnaire will be used to determine how daily pain levels change throughout the study. Three questions assess current pain, worst pain in past 7 days, and worse pain in past month. These three questions are separately assessed for pain.
Brief Pain Inventory Scale (BPI) | Up to 32 weeks
  The BPI is a 15-item self-report measure of pain intensity and pain interference with daily life. The Brief Pain Inventory (BPI) is scored separately for its two main sections: Pain Severity and Pain Interference. It includes questions about the intensity of pain at its "worst," "least," "average," and "right now" over the past week. Respondents rate the severity of pain on a numeric rating scale (NRS) from 0 to 10. The Pain Interference section evaluates the extent to which pain interferes with various aspects of the individual's life. The Pain Severity Score is calculated with the average score of the four items assessing pain severity. This average represents the overall pain severity experienced by the individual. This questionnaire will be used to determine how current pain levels change throughout the study.
Life Satisfaction Questionnaire (LiSAT) | Up to 32 weeks
  The LiSAT is a self-report instrument used to assess overall satisfaction with various life domains. It provides a comprehensive assessment of life satisfaction.
  The LiSAT consists of items that assess satisfaction across several domains of life, such as:
  work, leisure activities and free time, economy, relationships with friends, relationships with relatives, sexual life/partner relationship, physical health, psychological health, and safety.
  Respondents rate their satisfaction within each domain using a Likert-type scale, with response options ranging from "very dissatisfied" to "very satisfied".
  Each response is assigned a numerical value. After completing the questionnaire, scores for each domain are summed or averaged to obtain a total score or subscale scores representing satisfaction within specific life domains. Higher scores indicate greater satisfaction within the respective domain.
Post-traumatic Stress Disorder Checklist (PCL-5) | Up to 32 weeks
  The PTSD Checklist (PCL-5) is a widely used self-report measure used to assess symptoms of post-traumatic stress disorder (PTSD). It consists of 20 items that correspond to the Diagnostic and Statistical criteria for PTSD. Respondents rate the frequency of symptoms over the past month on a scale from 0 (Not at all) to 4 (Extremely). There are different cutoff scores used for diagnosing PTSD or assessing the severity of symptoms, but higher total scores generally indicate more severe PTSD symptoms.
  * 0-31: Subclinical range (minimal to no PTSD symptoms)
  * 32-37: Mild PTSD symptoms
  * 38-43: Moderate PTSD symptoms
  * 44 and above: Severe PTSD symptoms
The Patient-Reported Outcomes Measurement Information System (PROMIS 29+2) | Up to 32 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS 29+2) profile is a comprehensive assessment tool used to evaluate various aspects of health-related quality of life (HRQOL) across physical, mental, and social domains.
  Respondents rate their experiences over the past 7 days using a Likert-type scale, with response options ranging from 1 to 5. Higher scores indicate greater impairment or severity of symptoms, depending on the specific domain being assessed.
  For scoring, each item is scored based on the response provided by the respondent. Scores for items within each domain are aggregated to calculate domain scores. The questionnaire provides individual scores for each domain assessed, allowing for a comprehensive profile of the respondent's health-related quality of life. Total for each domain is assessed. Higher scores typically indicate greater impairment or symptom severity, while lower scores indicate better functioning or fewer symptoms.
Patient Health Questionnaire-9 (PHQ-9) | Up to 32 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used screening tool for depression. It consists of nine questions that ask about symptoms experienced over the past two weeks. Each question is scored on a scale from 0 to 3, with responses ranging from "not at all" to "nearly every day."
  To score the PHQ-9:
  1. Assign a score from 0 to 3 for each question based on the response:
     * "Not at all" = 0
     * "Several days" = 1
     * "More than half the days" = 2
     * "Nearly every day" = 3
  2. Sum the scores for all nine questions to obtain a total score, which can range from 0 to 27.
  Interpretation of the total PHQ-9 score is as follows:
  * 0-4: Minimal depression symptoms
  * 5-9: Mild depression symptoms
  * 10-14: Moderate depression symptoms
  * 15-19: Moderately severe depression symptoms
  * 20-27: Severe depression symptoms
Generalized Anxiety Disorder Scale | Up to 32 weeks
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a widely used screening tool designed to assess the severity of generalized anxiety disorder (GAD) symptoms. It consists of seven questions that ask about symptoms experienced over the past two weeks. Each question is scored on a scale from 0 to 3, with responses ranging from "not at all" to "nearly every day." To score the GAD-7 questions are rated from 0 to 3.
  * "Not at all" = 0
  * "Several days" = 1
  * "More than half the days" = 2
  * "Nearly every day" = 3 The sum of the scores for all seven questions obtain a total score, which can range from 0 to 21.
  Interpretation of the total GAD-7 score is as follows:
  * 0-4: Minimal anxiety symptoms
  * 5-9: Mild anxiety symptoms
  * 10-14: Moderate anxiety symptoms
  * 15-21: Severe anxiety symptoms

SECONDARY OUTCOMES:
Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) Tool | Up to 32 weeks
  The Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) tool is a comprehensive screening instrument used to assess an individual's substance use across multiple categories. It's designed to provide a thorough evaluation of substance use behaviors, including tobacco, alcohol, prescription medications, and other substances.
Richmond Agitation-Sedation Scale (RASS) | Up to 26 weeks
  The Richmond Agitation-Sedation Scale (RASS) measures a patient's agitation or sedation level.
  The scale ranges from -5 to +4:
  Based on the observed behavior, assign a numerical score on the RASS scale:
  * +4: Combative, violent, immediate danger to staff
  * +3: Very agitated, pulling at tubes, aggressive
  * +2: Agitated, restless, anxious, attempting to sit up
  * +1: Restless, uneasy, fidgety, tense
  * 0: Alert and calm
  * -1: Drowsy, not fully alert but able to be aroused
  * -2: Light sedation, easily aroused, briefly following commands
  * -3: Moderate sedation, difficult to arouse but responds to stimuli
  * -4: Deep sedation, minimal or no response to stimuli
  * -5: Unarousable, no response to stimuli
Clinician-Administered Dissociative States Scale (CADSS) | Up to 26 weeks
  The CADSS is a tool used to assess dissociative states induced by drugs or other factors. The Clinician-Administered Dissociative States Scale (CADSS) is used to measure the severity of dissociative states induced by drugs or other factors. Each item on the scale is rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (extremely). The total score is calculated by summing up the scores for all items on the scale.To score the CADSS, each item is rated on a 5-point Likert scale (0 to 4) based on the severity of the symptom described. The total score is summed for all 23 items to obtain the total CADSS score. This total score ranges from 0 to 92, with higher scores indicating greater severity of dissociative symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

REFERENCES:
- [Background] Urits I, Jung JW, Amgalan A, Fortier L, Anya A, Wesp B, Orhurhu V, Cornett EM, Kaye AD, Imani F, Varrassi G, Liu H, Viswanath O. Utilization of Magnesium for the Treatment of Chronic Pain. Anesth Pain Med. 2021 Feb 6;11(1):e112348. doi: 10.5812/aapm.112348. eCollection 2021 Feb. PMID 34221945
- [Background] Orhurhu V, Orhurhu MS, Bhatia A, Cohen SP. Ketamine Infusions for Chronic Pain: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Anesth Analg. 2019 Jul;129(1):241-254. doi: 10.1213/ANE.0000000000004185. PMID 31082965